CLINICAL TRIAL: NCT01277354
Title: Effectiveness of Cognitive Processing Therapy in Reducing Post-traumatic Symptoms and Enhancing Birth Outcomes in Pregnant Women With a Previous Pregnancy Loss or Complication
Brief Title: Effectiveness of Cognitive Processing Therapy in Pregnant Women With a History of Pregnancy Loss/Complication
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding
Sponsor: University of Pennsylvania (Other)
Collaborators: March of Dimes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 810277; March of Dimes Foundation (Other Grant/Funding Number: 12-FY07-679)
Record Dates: First submitted 2010-11-29; First posted 2011-01-14 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Post-traumatic Stress Disorder; Stress Disorders; Anxiety; Depression
Keywords: Cognitive Processing Therapy (CPT)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Processing Therapy (Active Comparator): Participants are seen weekly for six weeks for therapy. At visits 2, 4, and 6 they also complete ratings.
  Interventions: Behavioral: Cognitive Processing Therapy
- Waitlist (Placebo Comparator): Participants come in at the end of weeks 2, 4, and 6 to complete ratings but do not receive therapy.
  Interventions: Behavioral: Waitlist Placebo

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — CPT utilizes a combination of a) exposure therapy aimed at extinguishing fear and distress induced by memories and external cues associated with the trauma, and b) cognitive behavioral techniques that address faulty thinking patterns developed to promote a sense of control over possible future traumas, but that instead perpetuate PTSD symptoms. In CPT, exposure to the traumatic memory occurs through writing and reading for periods of time determined by the client and is confined to the week of the 4th and 5th sessions. These sessions are otherwise used to identify "stuck-points", i.e., distorted interpretations regarding the trauma and unrealistic beliefs regarding self and others.
  Arms: Cognitive Processing Therapy
Behavioral: Waitlist Placebo — Behavioral ratings are conducted by a blind rater.
  Arms: Waitlist

SUMMARY:
The purpose of this study is to examine the effects of experiencing a previous pregnancy loss or complication on current physiological and emotional aspects of a current pregnancy.

DETAILED DESCRIPTION:
This study will assess the effectiveness of cognitive processing therapy (CPT) or cognitive behavioral therapy (CBT) among women who are experiencing symptoms of post-traumatic stress disorder (PTSD) and/or anxiety relating to a previous pregnancy loss or complication. Lastly, this study includes an option to participate in a procedure whereas startle response will be measured using the eyeblink reflex twice during pregnancy and once in the postpartum period. Startle response is examined using a standard acoustic startle procedure whereby heart rate, skin temperature and eye blinking reflex are measured.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) criteria for full PTSD or partial PTSD.
* Clinician Administered PTSD Scale (CAPS) score of ≥18.
* Gestational age at the time of presentation is between 8 and 30 weeks.
* History of at least one of the following: previous pregnancy loss or losses, voluntary termination due to fetal anomaly, obstetrical complication including childbirth, premature birth (<32 weeks), unexpected neonatal complication, emergency C-section, neonatal death within 28 days of delivery.
* Fluency in spoken and written English.

Exclusion Criteria:

* Presence of any lifetime or comorbid DSM-IV Axis I psychotic disorder (including bipolar disorder and MDD (Major Depressive Disorder) with psychotic features and excepting Psychosis NOS (Not Otherwise Specified) related to sensory hallucinations, i.e. reexperiencing symptoms).
* Presence of any comorbid Axis I or Axis II (as determined using the SCID-II (Structured Clinical Interview for DSM-IV)) disorder, which would require immediate treatment or renders the subject clinically unsuitable for this RTC (randomized clinical trial).
* History of PTSD due to a NON-Pregnancy related traumatic event.
* Presence of a known abnormality in the present fetus.
* Presence of a serious medical or neurological illness.
* Starting a new psychotropic agent within the previous 3 months.
* Assessed to require a new psychotropic medication at the screening appointment or an adjustment in current dose of psychotropic medication.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Neill Epperson, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Center for Women's Behavioral Wellness, University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Forray A, Mayes LC, Magriples U, Epperson CN. Prevalence of post-traumatic stress disorder in pregnant women with prior pregnancy complications. J Matern Fetal Neonatal Med. 2009 Jun;22(6):522-7. doi: 10.1080/14767050902801686. PMID 19488936
- See also: Program Website — http://www.med.upenn.edu/womenswellness/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this project was slow and only two subjects matriculated during the period that this project was active.
Groups:
- CPT Group: Participants are seen weekly for six weeks for therapy. At visits 2, 4, and 6 they also complete ratings.
- Waitlist Group: Participants come in at the end of weeks 2, 4, and 6 to complete ratings but do not receive therapy.
Period: Overall Study
Arm/Group | CPT Group | Waitlist Group
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPT Group | Waitlist Group | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: CPT Effectiveness as Determined by the Number of Participants With CAPS Score Decrease of 50% From Baseline to Week 6
Description: The CAPS will be used in the diagnosis of PTSD, assessment of the impact of symptoms on function, assessment of the severity of symptoms at baseline, and weekly throughout the study. The CAPS in this particular study must decrease by 50% for CPT to be deemed effective.
Time Frame: 6 weeks
Population: Please note that there were only a total of 2 participants involved in this study. Funding was lost to continue and the study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | CPT Group | Waitlist Group
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Through study completion
Arm/Group | CPT Group | Waitlist Group
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
The limitations of this trial include an insufficient number of subjects enrolled which prohibits our ability to analyze the data in any meaningful fashion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No